CLINICAL TRIAL: NCT05603429
Title: Investigation of Myocardial Protection Level by Oxidative Stress and Endothelial Damage With Two Cardioplegia Methods Used During Cardiac Surgery
Brief Title: Investigation of Myocardial Protection Level With Specific Cardioplegia Methods in Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Dr. Siyami Ersek Thoracic and Cardiovascular Surgery Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Fatih KIZILYEL, Principal Investigator, Dr. Siyami Ersek Thoracic and Cardiovascular Surgery Training and Research Hospital
Other Study IDs: HNEAH-KAEK 2022/43-3507
Record Dates: First submitted 2022-03-11; First posted 2022-11-02 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Bypass Complication; Cardioplegia Solution Adverse Reaction; Endothelial Degeneration; Oxidative Stress; Aortic Valve Stenosis; Coronary Artery Disease
Keywords: Coronary Artery Bypass Grafting; Cardioplegia; Cardiopulmonary Bypass; Aortic Valve Replacement; Endothelial Damage; Oxidative Stress
MeSH Terms: conditions — Aortic Valve Stenosis; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Biospecimen Retention: Samples Without DNA — Venous blood specimens taken from peripheral venous cannula and retrograde cardioplegia cannula
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- CABG with cold blood cardioplegia: Subjects undergo Elective Coronary Artery Bypass Grafting with the use of cold blood cardioplegia solution for myocardial protection
  Interventions: Diagnostic Test: Endocan, E-Selectin, TNF-alpha, Total Oxidant and Antioxidant Status
- CABG with Del Nido: Subjects undergo Elective Coronary Artery Bypass Grafting with the use of Del Nido cardioplegia solution as myocardial protection
  Interventions: Diagnostic Test: Endocan, E-Selectin, TNF-alpha, Total Oxidant and Antioxidant Status
- AVR with cold blood cardioplegia: Subjects undergo Aortic Valve Replacement with the use of cold blood cardioplegia solution as myocardial protection
  Interventions: Diagnostic Test: Endocan, E-Selectin, TNF-alpha, Total Oxidant and Antioxidant Status
- AVR with Del Nido: Subjects undergo Aortic Valve Replacement with the use of Del Nido cardioplegia solution as myocardial protection
  Interventions: Diagnostic Test: Endocan, E-Selectin, TNF-alpha, Total Oxidant and Antioxidant Status

INTERVENTIONS:
Diagnostic Test: Endocan, E-Selectin, TNF-alpha, Total Oxidant and Antioxidant Status — Endocan, E-Selectin, TNF-alpha, Total Oxidant and Antioxidant Status measurements for determining Endothelial Damage and Oxidative Stress

SUMMARY:
Investigating the myocardial effects of cold blood cardioplegia and del nido cardioplegia solution, which are routinely used in clinical practice, will contribute to the studies in the literature on the safety and efficacy of these two methods.

For this purpose, patients with coronary artery disease that going to be Coronary Artery Bypass Graft (CABG) surgery will be classified within the scope of the SYNTAX score, the level of exposure to cardioplegia change in proportion to their score will be examined. Also, left ventricular muscle mass will be calculated in patients who will undergo Aortic Valve replacement (AVR) due to Aortic Stenosis, and myocardial protection level proportional to muscle mass will be examined, and cardioplegia efficiency will be compared.

DETAILED DESCRIPTION:
Endocan, E-Selectin, TNF(Tumor Necrosis Factor)-alpha, Total Oxidant and Antioxidant status will be studied on sequential blood samples taken from patients who will undergo Elective Coronary Artery Bypass Grafting operation and aortic valve replacement, via retrograde cardioplegia cannula before induction, at the beginning of cardiopulmonary bypass and after removing the cross-clamp. With routinely used parameters like hemogram, lactate, liver and kidney function tests morbidity-mortality rates for specific cardioplegia technique will be compared

ELIGIBILITY:
Inclusion Criteria:

* Subjects planned to have elective coronary artery bypass grafting for coronary artery disease
* Subjects planned to have elective aortic valve surgery due to aortic valve stenosis
* Patients aged 18-75 years
* BMI of 18.5-30
* Diabetic and non-diabetic patients
* Smokers and non-smokers

Exclusion Criteria:

* Subjects under 18 years old
* Subjects older than 75 years
* Patients requiring valve surgery with coronary artery bypass
* Patients requiring aortic valve surgery with pathologies other than aortic valve stenosis
* Patients requiring mitral or tricuspid valve surgery
* Patients undergoing emergency coronary bypass
* BMI > 30 obese patients

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with coronary artery disease and aortic valve stenosis irrespectively
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2022-10-13 (Actual); Primary Completion 2023-07-25 (Actual); Study Completion 2023-08-08 (Actual)

PRIMARY OUTCOMES:
Del Nido has beneficial effect for Endothelial function | through study completion, an average of 1 year
  Two groups with the protection of Del Nido cardioplegia solution, might have lesser Adverse outcomes from cardiopulmonary bypass and cross-clamping irrespectively, with measurements of BLOOD ENDOCAN (ng/ml) and E-SELECTIN LEVELS measured from venous blood specimens.
  Endocan and E-selectin levels to be measured by ELISA (ng/ml), expected to be much higher in the blood cardioplegia group because of the protective affect of Del nido cardioplegia.
  The venous blood specimens are going to be collected on different operation phases; after cannulation just before the beginning of cardiopulmonary bypass, after removing the cross-clamp before decannulation
Del Nido cardioplegia solution has lesser oxidative effect comparing to blood cardioplegia | through study completion, an average of 1 year
  Two groups with the protection of Del Nido cardioplegia solution, expected to be lesser oxidative affect with comparing of the TOTAL OXIDANT AND ANTIOXIDANT STATUS measured with specific assay kits from venous blood specimens First venous blood specimen will be taken from peripheral blood, 2nd and 3rd will be taken from coronary sinus blood through retrograde cardioplegia cannula; The venous blood specimens are going to be collected on different operation phases: 1st; after cannulation just before the beginning of cardiopulmonary bypass, 2nd; after removing the cross-clamp before decannulation
SYNTAX effect (SYNergy between PCI{Percutaneous Coronary Intervention} with TAXUS and Cardiac. Surgery) | through study completion, an average of 1 year
  The SYNTAX score has the potential to grade coronary anatomy and to guide patient selection toward the optimal revascularisation treatment to treat complex coronary artery disease (CAD).
  Subjects with Coronary Artery Disease might have proportional outcomes with SYNTAX score of individuals based upon parameters measured from venous blood specimens That means one wiht the higher SYNTAX score, expected to have higher difference in the blood cardioplegia group compared to Del Nido cardioplegia group because of the lesser protective affects to the myocardium. (ENDOCAN, E-SELECTIN, TOTAL OXIDANT AND ANTIOXIDANT STATUS measured by specific assay kits)
LVMI effect | through study completion, an average of 1 year
  In patients with severe symptomatic Aortic stenosis, concentric left ventricular(LV) geometry and severe LV hypertrophy by echocardiography have been associated with increased mortality after aortic valve replacement. So, demonstration of the relation of LV mass with myocardial protection levels might be important in the aortic stenosis patients for postoperative morbidity and mortality.
  Subjects with Aortic Valve Stenosis might have proportional outcomes with Left Ventricular Mass Index (LVMI) of individuals based upon parameters measured from venous blood specimens. (ENDOCAN, E-SELECTIN, TOTAL OXIDANT AND ANTIOXIDANT STATUS measured by specific assay kits)

CONTACTS AND LOCATIONS:
Overall Officials: Bulend KETENCI, Study Chair — Dr. Siyami Ersek Thoracic and Cardiovascular Surgery Training and Research Hospital
Locations (1):
- Dr. Siyami Ersek Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Li Y, Lin H, Zhao Y, Li Z, Liu D, Wu X, Ji B, Gao B. Del Nido Cardioplegia for Myocardial Protection in Adult Cardiac Surgery: A Systematic Review and Meta-Analysis. ASAIO J. 2018 May/Jun;64(3):360-367. doi: 10.1097/MAT.0000000000000652. PMID 28863040
- [Background] O'Blenes SB, Friesen CH, Ali A, Howlett S. Protecting the aged heart during cardiac surgery: the potential benefits of del Nido cardioplegia. J Thorac Cardiovasc Surg. 2011 Mar;141(3):762-70. doi: 10.1016/j.jtcvs.2010.06.004. Epub 2010 Jul 24. PMID 20656301
- [Background] Ad N, Holmes SD, Massimiano PS, Rongione AJ, Fornaresio LM, Fitzgerald D. The use of del Nido cardioplegia in adult cardiac surgery: A prospective randomized trial. J Thorac Cardiovasc Surg. 2018 Mar;155(3):1011-1018. doi: 10.1016/j.jtcvs.2017.09.146. Epub 2017 Nov 13. PMID 29246552
- [Result] Orak Y, Kocarslan A, Boran OF, Acipayam M, Eroglu E, Kirisci M, Doganer A. Comparison of the operative and postoperative effects of del Nido and blood cardioplegia solutions in cardiopulmonary bypass surgery. Braz J Cardiovasc Surg. 2020 Oct 1;35(5):689-696. doi: 10.21470/1678-9741-2019-0436. PMID 33118734